CLINICAL TRIAL: NCT05702489
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2/3 Study to Evaluate the Efficacy and Safety of ZX-7101A Tablets in Adults with Uncomplicated Influenza
Brief Title: A Study to Evaluate the Efficacy and Safety of ZX-7101A Tablets in Adults with Uncomplicated Influenza
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX-7101A-202
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ZX-7101A low dose group (Experimental): 40 mg, tablet, single oral administration when the subject screened successfully
  Interventions: Drug: ZX-7101A
- ZX-7101A high dose group (Experimental): 80 mg, tablet, single oral adminitration when the subject screened successfully
  Interventions: Drug: ZX-7101A
- Placebo control (Placebo Comparator): Analog tablet with no active ingredient, single oral administration when the subject screened successfully
  Interventions: Drug: ZX-7101A

INTERVENTIONS:
Drug: ZX-7101A — a drug to treatment influenza in Chinese adults

SUMMARY:
The goal of this clinical trial is to compare ZX-7101A in Chinese Adults patients with uncomplicated influenza. The main questions it aims to answer are:

* The efficacy of ZX-7101A in Chinese Adults patients with uncomplicated influenza.
* The safety of ZX-7101A in Chinese Adults patients with uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 to ≤64 years of age at the time of signing the ICF.
* Patients in the screening period met the following criteria: (1) rapid influenza diagnostic test (RIDT) or polymerase chain reaction (PCR) test positive; (2) fever ≥ 37.3℃ (axillary temperature) at screening; if taking antipyretics, axillary temperature ≥ 37.3℃ after taking the drug (more than 4 hours). (3) At least one of flu-related systemic symptoms is moderate or greater in severity: a. muscle or joint pain, b. fatigue, c. headache, d. fever. (4) At least one of the influenza-related respiratory symptoms is moderate or greater in severity: a. nasal congestion, b. sore throat, c. cough.
* The first occurrence of influenza symptoms ≤ 48 hours from the time of patient randomization.

Exclusion Criteria:

* Patients with influenza virus infection requiring hospitalization.
* High-risk population.
* Bronchitis, pneumonia, pleural effusion or interstitial disease suspected by a clinician or confirmed by chest imaging [X-ray (anteroposterior or anteroposterior)/CT] and judged clinically significant by the investigator at screening.
* Patients who have developed acute respiratory tract infection, otitis media, and sinusitis within 2 weeks before screening.
* Patients with other infections requiring systemic anti-infective treatment, or blood routine examination at screening: white blood cell count (WBC) > 10.0 × 109/L.
* Patients with purulent sputum or suppurative tonsillitis.
* Those who have difficulty in swallowing drugs or have a history of gastrointestinal diseases that seriously affect drug absorption.
* Medications against influenza virus within 7 days prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
The time to the remission of all influenza symptoms (hours) | from accepting ZX-7101A until the 15 days after the first dosing
  Defined as the time from the start of study treatment to the time all flu symptoms are relieved. Symptom relief was defined as all seven influenza symptoms assessed by the subject on the subject diary card(Stuffy nose, sore throat, cough, muscle or joint pain, fatigue, headache, fever or chills/sweating) were 0 (asymptomatic) or 1 (mild);

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | from accepting ZX-7101A until the 15 days after the first dosing
  The Number of Participants with Treatment-Related Adverse Event will be evalated as the change of vital signs, electrocardiogram (P Wave, QRS Complex, QT Interval), physical examination, and Laboratory test compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: hong wen Zhang, doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No